CLINICAL TRIAL: NCT03791385
Title: Effectiveness of Picture Exchange Communication System (PECS) on Dental Plaque and Gingival Health of Children With Autism
Brief Title: Effectiveness of Picture Exchange Communication System on Gingival Health of Children With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20110011
Record Dates: First submitted 2018-12-23; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Picture Exchange Communication System (PECS); Tooth-brushing program; Gingival index; Plaque index
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Children with ASD ages 4-16 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study subjects (Experimental): Children with ASD and their parents/caregivers were trained on tooth-brushing twice, two weeks apart using Picture Exchange Communication System (PECS) PECS as a pictures/cards series showing a structured tooth-brushing method.
  Interventions: Behavioral: Picture Exchange Communication System (PECS)

INTERVENTIONS:
Behavioral: Picture Exchange Communication System (PECS) — A communication system frequently used with non-verbal children with autism spectrum disorders (ASD) that uses a series of pictures that describe how a certain activity is done, in our case showing a structured method and technique for teeth brushing.

SUMMARY:
The Picture Exchange Communication System (PECS) is a communication system for children with autism spectrum disorders (ASD). The aim of this study was to assess the effect of a PECS-based tooth-brushing program on gingival health in children with ASD and assess parents' perception of PECS. This was a prospective interventional study. Using PECS as a pictures/cards series showing a structured tooth-brushing method, 37 children with ASD (31 males, 6 females) (average age 9.49±4.10, 4-16 years) and their parents/caregivers were trained on tooth-brushing twice, two weeks apart. Data collected after examinations (baseline, 3, 6-months) included gingival and plaque indices (GI, PI) and two questionnaires (baseline, 6-months) for demographic data and parents' perception of PECS including: difficulty rating (easy, hard, very hard) and PECS usefulness.

DETAILED DESCRIPTION:
The need for improved oral hygiene routines in individuals with autism spectrum disorders (ASD) has been documented in many reports. The Picture Exchange Communication System (PECS), which is a series of pictures that show a structured method and technique for teeth brushing, was chosen for this study since it is a proven communication system for children with autism spectrum disorders (ASD).

The aim of the study was to assess the effect of a PECS-based tooth-brushing program on gingival health in children with ASD and assess parents' perception of PECS.

This was a prospective interventional study. Using PECS as a pictures/cards series showing a structured tooth-brushing method, 37 children with ASD (31 males, 6 females) (average age 9.49±4.10, 4-16 years) and their parents/caregivers were trained on tooth-brushing twice, two weeks apart. The pictures were placed in the bathroom, at home and/or at the autism center. Data collected after examinations (baseline, 3, 6-months) included gingival and plaque indices (GI, PI) and two questionnaires (baseline, 6-months) for demographic data and parents' perception of PECS including: difficulty rating (easy, hard, very hard) and whether they found PECS useful in teaching their children how to brush their teeth (yes or no).

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with ASD.
* Age between 4 and 18 years old.

Exclusion Criteria:

* Children unable to cooperate for data collection (poor behavior during dental examination).

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Gingival index score | 6 months
  This score indicates the level of gingival inflammation upon examination of teeth, reported as the average score calculated as (total score for all teeth/number of examined teeth): Score 0 (Absence of inflammation), Score 1 (Mild inflammation: slight change in colour (more red) and little change in texture (loss of stippling), No bleeding on probing), Score 2 (Moderate inflammation: moderate glazing, redness, edema and hypertrophy; bleeding on probing), Score 3 (Severe inflammation: marked redness and edema; tendency to spontaneous bleeding; ulceration). A lower score indicates less gingival inflammation (better gingival health) and vice versa.
Plaque index score | 6 months
  This score indicates the level of plaque (and reflects level of oral hygiene) upon examination of teeth, reported as the average score, calculated as (total score for all teeth/number of examined teeth): Score 0 (No plaque), Score 1 (Plaque not visible by eye, only detectable using a dental probe), Score 2 (Plaque visible by eye & detectable with a dental probe along the gingival margin of the tooth), Score 4 (Thick layer of plaque visible by eye & detectable by probe covering more than the gingival margin of the tooth). A lower score indicates less plaque (meaning better oral hygiene) and vice versa.

SECONDARY OUTCOMES:
Parents' rating of PECS difficulty | 6 months
  Parents were asked to rate PECS difficulty as: easy, hard, very hard. This was assessed through a questionnaire.
PECS usefulness | 6 months
  Parents were asked whether PECS was useful in teaching their children how to brush their teeth: yes, no. This was assessed through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ola B Al-Batayneh, Study Director — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

REFERENCES:
- [Background] Pilebro C, Backman B. Teaching oral hygiene to children with autism. Int J Paediatr Dent. 2005 Jan;15(1):1-9. doi: 10.1111/j.1365-263X.2005.00589.x. PMID 15663439
- [Background] Charlop-Christy MH, Carpenter M, Le L, LeBlanc LA, Kellet K. Using the picture exchange communication system (PECS) with children with autism: assessment of PECS acquisition, speech, social-communicative behavior, and problem behavior. J Appl Behav Anal. 2002 Fall;35(3):213-31. doi: 10.1901/jaba.2002.35-213. PMID 12365736
- [Background] Lerna A, Esposito D, Conson M, Massagli A. Long-term effects of PECS on social-communicative skills of children with autism spectrum disorders: a follow-up study. Int J Lang Commun Disord. 2014 Jul-Aug;49(4):478-85. doi: 10.1111/1460-6984.12079. Epub 2014 Mar 21. PMID 24655345
- [Background] Eslami N, Movahed T, Asadi M. Parents' Perceptions of the Oral Health-related Quality of Life of their Autistic Children in Iran. J Clin Pediatr Dent. 2018;42(6):422-426. doi: 10.17796/1053-4625-42.6.3. Epub 2018 Aug 7. PMID 30085870